CLINICAL TRIAL: NCT02487654
Title: Ectopy Triggering Ganglionated Plexus Ablation to Prevent Atrial Fibrillation
Acronym: GANGLIA-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13SM0713
Record Dates: First submitted 2013-11-25; First posted 2015-07-01 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal atrial fibrillation; Pulmonary vein isolation; Ganglionated plexus; Radiofrequency ablation; Pulmonary vein ectopy; High frequency stimulation; autonomic nervous system; Ganglionated plexi; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation (Active Comparator): Conventional endocardial radiofrequency catheter ablation for pulmonary vein isolation.
  Interventions: Procedure: Pulmonary vein isolation
- Ganglionated plexus ablation (Experimental): Endocardial radiofrequency catheter ablation of ganglionated plexus in the left atrium
  Interventions: Procedure: Ganglionated plexus ablation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Conventional endocardial radiofrequency catheter ablation for pulmonary vein isolation.
  Other Names: PVI
  Arms: Pulmonary vein isolation
Procedure: Ganglionated plexus ablation — Endocardial radiofrequency catheter ablation of ganglionated plexus in the left atrium
  Other Names: GP ablation
  Arms: Ganglionated plexus ablation

SUMMARY:
Atrial fibrillation (AF) is a common heart rhythm disorder which can significantly affect a patient's quality of life and cause strokes. Abnormal electrical activity from the pulmonary veins are thought to be the most common cause of this condition. Current ablative strategy in drug refractory AF is pulmonary vein isolation (PVI), where the pulmonary veins are electrically isolated from the body of the left atrium. However, success rate of this procedure remain ~50-70% for a single procedure despite advances in mapping and ablation techniques.

Ganglionated plexuses (GP) are dense clusters of nerves in the atria that are implicated in AF. Endocardial high frequency stimulation (HFS) delivered within the local atrial refractory period can trigger ectopy and AF from specific GP sites (ET-GP). The aim of this study was to understand the role of ET-GP ablation in the treatment of AF by comparing two different strategies:

1. Pulmonary vein isolation alone
2. GP ablation alone

DETAILED DESCRIPTION:
This is a prospective, multi-centre study recruiting patients with paroxysmal AF indicated for AF ablation.

180 patients will be recruited. Patients are randomised to either GP ablation alone or to PVI. All antiarrhythmics are stopped for at least 48 hours prior to their procedures.

All have general anaesthesia and CARTO system (Biosense Webster, inc.) are used for 3D electroanatomical mapping of the left atrium.

Patients randomised to GP ablation will have high frequency mapping performed within the atrial refractory period to identify ectopy or AF triggering GP (ET-GP) sites in the left atrium. Patients in this group will only have GP ablation and will not have pulmonary veins isolated.

The primary endpoint is any documented atrial arrhythmia 30 seconds or more after a 3 month blanking period. This will be assessed for up to 12 months post-procedure, using 48hr Holter monitors at 3, 6, 9 and 12 month intervals.

Secondary endpoints include mortality, major complications and redo procedures.

ELIGIBILITY:
Inclusion Criteria:

* Males or females eighteen (18) to eighty five (85) years old
* Paroxysmal atrial fibrillation
* Suitable candidate for catheter ablation
* Signed informed consent

Exclusion Criteria:

* Contraindication to catheter ablation
* Presence of a cardiac thrombus
* valvular disease that is grade moderate or greater
* Any form of cardiomyopathy
* On amiodarone therapy
* Severe cerebrovascular disease
* Active gastrointestinal bleeding
* Renal failure (on dialysis or at risk of requiring dialysis)
* Active infection or fever
* Life expectancy shorter than the duration of the trial
* Allergy to contrast
* Intractable heart failure (NYHA Class IV)
* Bleeding or clotting disorders or inability to receive heparin
* Serum Creatinine >200umol/L
* Uncontrolled diabetes (HbA1c ≥73mmol/mol or HbA1c ≤64mmol/mol and Fasting Blood Glucose ≥9.2mmol/L)
* Malignancy needing therapy
* Pregnancy or women of childbearing potential not using a highly effective method of contraception
* Patients in current research or have recently been involved in any research prior to recruitment will not be included in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-10-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, PhD, Principal Investigator — Imperial College NHS Healthcare Trust
Locations (3):
- United Kingdom (3):
  - Hammersmith Hospital, London
  - St Bartholomew's Hospital, London
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Kim MY, Coyle C, Tomlinson DR, Sikkel MB, Sohaib A, Luther V, Leong KM, Malcolme-Lawes L, Low B, Sandler B, Lim E, Todd M, Fudge M, Wright IJ, Koa-Wing M, Ng FS, Qureshi NA, Whinnett ZI, Peters NS, Newcomb D, Wood C, Dhillon G, Hunter RJ, Lim PB, Linton NWF, Kanagaratnam P. Ectopy-triggering ganglionated plexuses ablation to prevent atrial fibrillation: GANGLIA-AF study. Heart Rhythm. 2022 Apr;19(4):516-524. doi: 10.1016/j.hrthm.2021.12.010. Epub 2021 Dec 13. PMID 34915187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrolement of participants was between 2017 and 2020
Period: Overall Study
Arm/Group | Pulmonary Vein Isolation | Ganglionated Plexus Ablation
Started | 53 | 63
Completed | 50 | 52
Not Completed | 3 | 11
Not completed — 4 withdrawndue to non-identifiable GPs during HFS mapping in the GPA group. | 0 | 4
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Vein Isolation | Ganglionated Plexus Ablation | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 64 (11) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 36 | 35 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With no Evidence of >30s Recurrent Atrial Arrhythmia Post-index Procedure
Description: That is documented recurrent atrial arrhythmia lasting 30 seconds or more after a blanking period of 3 months; the outcome measure will be assessed up to 12 months of follow-up with 48hr halter monitors arranged every 3 months to investigate Arrhythmia recurrence .
Time Frame: 3 to 12 months post-ablation.
Population: Number of patients with no evidence of Atrial arrhythmia recurrence, >30s, on a 48 hour Holter monitor during the initial 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Vein Isolation | Ganglionated Plexus Ablation
Number analyzed (Participants) | 50 | 52
Participants | 32 | 26
Statistical Analysis 1: Comparison: Pulmonary Vein Isolation vs Ganglionated Plexus Ablation; Test type: Superiority; p < 0.05, Log Rank

2. Secondary Outcome: Number of Participants Presenting a Reduction in the Usage of Antiarrhythmics Post-ablation
Description: The reduction was defined as either a decrease of dose or a cessation of a drug over a 12 month follow-up period post ablation.
Time Frame: 3 to 12 months post-ablation.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Vein Isolation | Ganglionated Plexus Ablation
Number analyzed (Participants) | 50 | 52
Participants | 12 | 16

3. Post Hoc Outcome: Extended Follow up to Assess Freedom From Atrial Arrhythmia Over a Prolonged Duration
Description: evidence of >30s atrial arrhythmia or symptoms consistent with arrhythmia recurrence, during routine clinical care, over an extended follow up period of 40 months.
Time Frame: 40 months post procedure.
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 12 months post procedure.
Arm/Group | Pulmonary Vein Isolation | Ganglionated Plexus Ablation
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/63
Other Adverse Events (participants affected / at risk) | 1/53 | 7/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pulmonary Vein Isolation (N=53) | Ganglionated Plexus Ablation (N=63)
Cardiac tamponade (Cardiac disorders) | 0 | 1 — Pericardiocentesis performed which successfully treated cardiac tamponade. No other complications, discharged following day of ablation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmonary Vein Isolation (N=53) | Ganglionated Plexus Ablation (N=63)
Pericarditis (Cardiac disorders) | 1 (1) | 7 (7) — Hospital attendance with symptoms consistent with pericarditis, conservatively managed with short course of analgesia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02487654/Prot_SAP_000.pdf